CLINICAL TRIAL: NCT04317443
Title: A Prospective Observational Comparison of Super-mini Percutaneous Nephrolithotomy (SMP) and Extracorporeal Shock Wave Lithotripsy (ESWL) for the Treatment of Renal Stones ≥20 mm in Children: An IAU Study
Brief Title: A Prospective Observational Comparison of SMP and ESWL for the Treatment of Renal Stones ≥20 mm in Children (IAU-04)
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: The International Alliance of Urolithiasis (Network)
Responsible Party: Sponsor
Other Study IDs: 2020-01
Record Dates: First submitted 2020-03-11; First posted 2020-03-23 (Actual); Last update posted 2020-04-30 (Actual); Status verified 2020-04

CONDITIONS: Kidney Stone
Keywords: percutaneous nephrolithotomy; pcnl; miniperc; smp; children
MeSH Terms: conditions — Kidney Calculi | interventions — Lithotripsy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Super-Mini Percutaneous Nephrolithotomy: Patients undergo SMP
  Interventions: Procedure: Super-mini percutaneous nephrolithotomy (SMP)
- Extracorporeal Shock Wave Lithotripsy: Patients undergo ESWL
  Interventions: Procedure: Extracorporeal Shock Wave Lithotripsy (ESWL)

INTERVENTIONS:
Procedure: Super-mini percutaneous nephrolithotomy (SMP) — SMP will be performed under general anesthesia in prone/supine position. Renal puncture will be performed under ultrasound/fluoroscopy guidance based on the preference of the participating surgeon. Tracts will be dilated to 14 Fr. Stone fragmentation will be performed with holmium laser and fragments will be extracted with the active suction system. For the exit strategy, placement of a nephrostomy tube or JJ stent will be decided by the participating surgeon.
  Groups: Super-Mini Percutaneous Nephrolithotomy
Procedure: Extracorporeal Shock Wave Lithotripsy (ESWL) — ESWL will be performed under sedation/analgesia, shock wave lithotripsy parameters will be determined based on the device and the settings of local center. For patients requiring multiple sessions, maximum 3 (or more) sessions will be allowed. Ureteral stenting prior to ESWL will be performed based on the decision of the participating center.
  Groups: Extracorporeal Shock Wave Lithotripsy

SUMMARY:
ESWL and PNL are the two treatment modalities for kidney stones greater than 20 mm in the pediatric population. ESWL is non-invasive, does not require anesthesia and inexpensive, but its success rate may be lower, and require multiple treatment sessions. On the contrary, PNL has a higher success rate, does not require multiple sessions but is an invasive method. Compared to standard PNL, miniaturized PNL systems have been shown to decrease complications with comparable success rates. SMP is a unique miniaturized PNL system with integrated active irrigation and suction systems. The current literature lacks studies comparing SMP and ESWL prospectively in the pediatric population. In this study, the effectiveness, reliability, and reusability of ESWL and SMP will be compared.

DETAILED DESCRIPTION:
To compare the success and complication rates of super-mini-percutaneous nephrolithotomy (SMP) and Extracorporeal Shock Wave Lithotripsy (ESWL) for the treatment of renal stones ≥20 mm in children.An international multicentre, prospective, observational study. Pediatric cases with renal Stones ≥20 mm who undergo ESWL or SMP will be evaluated and compared proespectively. The total number of departments planned to be included in the study is 10 and the number of cases is 180.

ELIGIBILITY:
Inclusion Criteria:

* Children ≤14 years old with renal Stones ≥20 mm
* Willing and able to sign informed consent
* Normal renal function
* No stone-related surgical history
* American Society of Anesthesiology (ASA) score 1-2

Exclusion Criteria:

* Congenital renal anomalies (horseshoe kidney, ureteropelvic junction obstruction)
* Uncorrected UTI
* Abnormal coagulation function
* Morbid obese children (BMI≥35）

Max Age: 14 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Pediatric patients undergoing SWL and SMP
Sampling Method: Probability Sample
Enrollment: 250 (Estimated)
Dates: Start 2020-05-01 (Estimated); Primary Completion 2021-05-01 (Estimated); Study Completion 2021-09-01 (Estimated)

PRIMARY OUTCOMES:
Stone free rate | 3-months
  Stone clearance on the computed tomography (2mm thickness)

SECONDARY OUTCOMES:
blood loss | Postoperative day 1
  Number of participants requiring blood transfusion after the procedure
auxiliary procedures | Postoperative month 3
  Number of patients requiring additional auxiliary procedures such as second look PCNL, SWL, Ureteroscopy
hospital stay | Postoperative month 3
  From date of admission until the date of discharge,length of hospital stay
complications | Postoperative month 3
  Rate of postoperative complications using the Clavien-Dindo system

IPD SHARING:
Plan to Share IPD: No